CLINICAL TRIAL: NCT00078273
Title: Indicated Prevention With At-Risk Gamblers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23848-C; R21MH067026 (NIH); DATR A2-AII
Record Dates: First submitted 2004-02-20; First posted 2004-02-24 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Gambling; Pathological Gambling; Problem Gambling
Keywords: Gambling; Pathological Gambling; Problem Gambling; College Students; Prevention
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Assessment Only Control (No Intervention): Completed Baseline and 6 month follow-up surveys only.
- Personalized Feedback Intervention (Experimental): See Intervention Description
  Interventions: Behavioral: Personalized Feedback Intervention
- Cognitive Behavioral Intervention (Experimental): See Intervention Description
  Interventions: Behavioral: Cognitive Behavioral Intervention

INTERVENTIONS:
Behavioral: Personalized Feedback Intervention — Sessions lasted for 60-90 minutes and used Motivational Interviewing (MI) to facilitate discussion of feedback from participants' survey responses. Sessions began with open-ended questions about contextual factors associated with participants' gambling, then review of each feedback section: gambling pattern; perceived gambling norms; positive expectancies and negative consequences of gambling; beliefs about control over gambling; and situational self-efficacy to avoid gambling. Participants were encouraged to consider the feedback in light of their personal goals. All participants received a copy of their feedback, a list of skills for limiting gambling and a resource/referral list.
  Arms: Personalized Feedback Intervention
Behavioral: Cognitive Behavioral Intervention — Participants completed either six weekly 1-hour sessions or attend four sessions containing the same content. Sessions covered functional analysis and gambling triggers; challenging cognitive distortions, with emphasis on illusions of control; coping with triggers; assertiveness; and relapse prevention. Participants received a pamphlet covering each week's topic (which was reviewed with the participant if a session was missed), as well as homework sheets and gambling diaries. CBI participants were asked to refrain from gambling for the duration of the group to provide an opportunity to practice and develop skills applicable to gambling and other behavior change situations.
  Arms: Cognitive Behavioral Intervention

SUMMARY:
The overall purpose of this study is to reduce the prevalence of gambling risk in college students by evaluating the effectiveness of different treatments in reducing gambling behavior and related negative consequences.

DETAILED DESCRIPTION:
Participants in this study will be randomly assigned to a personal feedback intervention (PFI) or assessment only for 3 years. The PFI intervention will be delivered in a single session. Measures will include the NORC DSM Screen for Problem Gambling (NODS), the South Oaks Gambling Screen (SOGS), Gambling Quantity and Perceived Norms, Perceived Injunctive Gambling Norms, Gambling Problems Index, gambling frequency, attitudes and beliefs about gambling and self-control, readiness to change, gambling expectancies, gambling motives, gambling risk perception, psychiatric symptoms, assertiveness, coping skills, substance use, alcohol-related problems, self-determination, and social desirability.

ELIGIBILITY:
Inclusion Criteria:

* College student
* South Oaks Gambling Screen (SOGS) score greater than 3

Exclusion Criteria:

* None, other than not meeting inclusion criteria

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2003-07; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
South Oaks Gambling Screen (SOGS) | 6-Months
  The 20-item South Oaks Gambling Screen (SOGS) measures gambling involvement and problem severity based on DSM-III-R pathological gambling criteria.
Gambling Quantity and Perceived Norms Scale (GQPN) | 6 Months
  The gambling quantity and perceived norms scale (GQPN) includes a six-item expenditure subscale assessing amount of money won/lost through gambling on a 10-point scale from $0 to more than $2000 over time-periods from the past month to past year. Additional items assess gambling frequency (on a 10-point scale from never to every day in the past year), disposable income (on an 11-point scale from less than $50 to more than $500 per month) and perceptions of gambling frequency and expenditure for the typical college student (perceived norms). Gambling expenditure was calculated as the expenditure subscale mean residualized on disposable income.
Gambling Frequency (SOGS) | 6 Months
  The SOGS was modified to assess internet gambling frequency and expand gambling frequency response options from a three- to a five-point scale with anchors of no times, one to 10 times, more than 10 times, less than weekly, weekly or more than weekly but less than daily, and daily. This modified frequency scale has been shown to correlate highly with other measures of gambling frequency.
Gambling Problems Index (GPI) | 6 Months
  Gambling problems (or negative consequences) were assessed using the 20-item Gambling Problems Index (GPI). Participants indicated how often, from never to more than 10 times in the past 6 months, they experienced consequences while, or as a result of, gambling.
National Opinion Research Center DSM-IV Screen for Pathological Gambling (NODS) | 6 Months
  DSM-IV [1] criteria for pathological gambling were assessed using the 17-item National Opinion Research Center DSM-IV Screen (NODS). Some criteria have multiple items, but possible scores range from 0-10 DSM-IV criteria endorsed in the past 6 months.

SECONDARY OUTCOMES:
Illusions of Control | 6 Months
  Illusions of control were assessed via a six-item subscale from the Beliefs About Control Scale (BACS), on a five-point scale ranging from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Larimer, Ph.D, Principal Investigator — University of Washington, Dept of Psychiatry & Behavioral Sciences
Locations (1):
- University of Washington; Department of Psychiatry and Behavioral Sciences, Seattle, Washington, United States

REFERENCES:
- [Result] Larimer ME, Neighbors C, Lostutter TW, Whiteside U, Cronce JM, Kaysen D, Walker DD. Brief motivational feedback and cognitive behavioral interventions for prevention of disordered gambling: a randomized clinical trial. Addiction. 2012 Jun;107(6):1148-58. doi: 10.1111/j.1360-0443.2011.03776.x. Epub 2012 Feb 28. PMID 22188239